CLINICAL TRIAL: NCT05484531
Title: A Multicentre, Prospective, Registry Study for Femtosecond Laser Corneal Lenticule Extraction for Advanced Refractive Correction (CLEAR) Procedure in Myopia and Astigmatism
Brief Title: CLEAR Procedure in Myopia and Astigmatism - Registry Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ziemer Ophthalmic Systems AG (Industry)
Responsible Party: Sponsor
Other Study IDs: CPFEM-0011-EU
Record Dates: First submitted 2022-07-29; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Myopia; Astigmatism
Keywords: CLEAR; Ziemer; FEMTO LDV; Astigmatism; Myopia; Lenticule extraction
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- CLEAR: Adult subjects suffering from myopia AND/OR astigmatism treated with CLEAR.
  Interventions: Device: CLEAR

INTERVENTIONS:
Device: CLEAR — Reduction or elimination of myopia from -0.50 D to -10.00 D, with astigmatism of 0 D to -5.00 D or without astigmatism, and MRSE of -0.50 D to -12.50 D in the eye to be treated in patients who are 18 years of age or older with documentation of stable manifest refraction over the past year as demonstrated by a change in sphere and cylinder of ≤ 0.50 D in magnitude

SUMMARY:
Multicenter, prospective, single-arm, observational, non-interventional post market clinical investigation (registry study) with the overall objective to assess safety and performance of CLEAR in a real world setting.

ELIGIBILITY:
Formal inclusion/exclusion criteria are not applicable to the study at hand, due to its observational and non-interventional nature.

Patients treated with the CLEAR application using FEMTO LDV Z8, enrolled in the study are expected not to present with any of the market-approved device's contraindications:

* Residual thickness of stromal bed that is less than 250 microns from the corneal endothelium
* Abnormal corneal topographic findings, e.g. keratoconus, pellucid marginal degeneration
* Ophthalmoscopic signs of progressive or unstable myopia or keratoconus (or keratoconus suspect)
* Irregular or unstable (distorted/not clear) corneal mires on central keratometry images
* Severe dry eye
* Active eye infection or inflammation
* Recent herpes eye infection or problems resulting from past infection
* Active autoimmune disease or connective tissue disease
* Uncontrolled diabetes
* High IOP fluctuations that are not controlled under medications and continuous visual field damage

Note 1: The above listed contraindications are a subject to change, as per PMS, risk management or other regulatory feedback, and will be covered and communicated to the participating investigators in the prospective updates of the Operator's Manual.

Note 2: Only eyes of patients treated bilaterally shall be included in the analysis covered by this registry study.

Note 3: Patient's targeted for "monovision" shall not be included in the analysis covered by this registry study.

Note 4: Clinical cases, that despite presenting any of the above listed contraindications, would still be enrolled in the study by the Investigator, may be subject to a sub-group statistical analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects (clients of the ophthalmology clinic) enrolled in several European countries, scheduled to undergo refractive surgery to correct myopia AND/OR astigmatic myopia.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
The percentage of eyes that achieve Uncorrected Distance Visual Acuity (UCDVA) of 20/40 (as per Snellen chart lines) or better | 1 day post surgery
  Uncorrected Distance Visual Accuity assessment
The percentage of eyes that achieve Uncorrected Distance Visual Acuity (UCDVA) of 20/40 (as per Snellen chart lines) or better | 1 month post surgery
  Uncorrected Distance Visual Accuity assessment
The percentage of eyes that achieve Uncorrected Distance Visual Acuity (UCDVA) of 20/40 (as per Snellen chart lines) or better | 3 months post surgery
  Uncorrected Distance Visual Accuity assessment
The percentage of eyes that achieve Uncorrected Distance Visual Acuity (UCDVA) of 20/40 (as per Snellen chart lines) or better | 6 months post surgery
  Uncorrected Distance Visual Accuity assessment
The percentage of eyes that achieve Uncorrected Distance Visual Acuity (UCDVA) of 20/40 (as per Snellen chart lines) or better | 12 months post surgery
  Uncorrected Distance Visual Accuity assessment

SECONDARY OUTCOMES:
Refractive target [D] | Preoperative assessment
  Expressed as MRSE
Corrected distance visual accuity (CDVA) | 1 day post surgery
  Values expressed as per Snellen Chart lines
Corrected distance visual accuity (CDVA) | 1 month post surgery
  Values expressed as per Snellen Chart lines
Corrected distance visual accuity (CDVA) | 3 months post surgery
  Values expressed as per Snellen Chart lines
Corrected distance visual accuity (CDVA) | 6 months post surgery
  Values expressed as per Snellen Chart lines
Corrected distance visual accuity (CDVA) | 12 months post surgery
  Values expressed as per Snellen Chart lines
Refraction [SphD, CylD, Axis] | 1 day post surgery
  Examination of both subjective and objective refraction.
  Values may be expressed as MRSE.
Refraction [SphD, CylD, Axis] | 1 month post surgery
  Examination of both subjective and objective refraction.
  Values may be expressed as MRSE.
Refraction [SphD, CylD, Axis] | 3 months post surgery
  Examination of both subjective and objective refraction.
  Values may be expressed as MRSE.
Refraction [SphD, CylD, Axis] | 6 months post surgery
  Examination of both subjective and objective refraction.
  Values may be expressed as MRSE.
Refraction [SphD, CylD, Axis] | 12 months post surgery
  Examination of both subjective and objective refraction.
  Values may be expressed as MRSE.
Assessment of changes in corneal topography [um] | Baseline and 1 month
  Following parameters will be assessed:
  * Simulated Keratometry (SimK) values
  * Average SimK (SimKavg)
  * Flat SimK (SimKf)
  * Steep SimK (SimKs)
  * Astigmatism [D, °]
  * Corneal anterior surface eccentricity
Assessment of changes in corneal topography [um] | Baseline and 3 months
  Following parameters will be assessed:
  * Simulated Keratometry (SimK) values
  * Average SimK (SimKavg)
  * Flat SimK (SimKf)
  * Steep SimK (SimKs)
  * Astigmatism [D, °]
  * Corneal anterior surface eccentricity
Assessment of changes in corneal topography [um] | Baseline and 6 months
  Following parameters will be assessed:
  * Simulated Keratometry (SimK) values
  * Average SimK (SimKavg)
  * Flat SimK (SimKf)
  * Steep SimK (SimKs)
  * Astigmatism [D, °]
  * Corneal anterior surface eccentricity
Assessment of changes in corneal topography [um] | Baseline and 12 months
  Following parameters will be assessed:
  * Simulated Keratometry (SimK) values
  * Average SimK (SimKavg)
  * Flat SimK (SimKf)
  * Steep SimK (SimKs)
  * Astigmatism [D, °]
  * Corneal anterior surface eccentricity
Assessment of changes in corneal pachymetry [um] | Baseline and 1 month
  Following parameters will be assessed:
  * Central corneal thickness [µm]
  * Thinnest corneal point [µm]
Assessment of changes in corneal pachymetry [um] | Baseline and 3 months
  Following parameters will be assessed:
  * Central corneal thickness [µm]
  * Thinnest corneal point [µm]
Assessment of changes in corneal pachymetry [um] | Baseline and 6 months
  Following parameters will be assessed:
  * Central corneal thickness [µm]
  * Thinnest corneal point [µm]
Assessment of changes in corneal pachymetry [um] | Baseline and 12 months
  Following parameters will be assessed:
  * Central corneal thickness [µm]
  * Thinnest corneal point [µm]
Assessment of changes in "white to white" [mm] | Baseline and 1 month
Assessment of changes in "white to white" [mm] | Baseline and 3 months
Assessment of changes in "white to white" [mm] | Baseline and 6 months
Assessment of changes in "white to white" [mm] | Baseline and 12 months
Number of Adverse Events observed in the study | Up to 12 months
  Following events will be recorded:
  * Adverse device effects (ADEs)
  * Surgical complications (intraoperative and post-operative)

IPD SHARING:
Plan to Share IPD: No